CLINICAL TRIAL: NCT04150042
Title: SHARON: Study of Metastatic Cancers in Patients Using Autologous Stems Cells and Potentiated Redox Cycling to Overcome Drug Resistance to Nitrogen Mustard Derivatives
Brief Title: SHARON: A Clinical Trial for Metastatic Cancer Using Chemotherapy and Patients' Own Stem Cells
Acronym: SHARON
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: General Oncology, Inc. (Industry)
Collaborators: Myriad Genetics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GO-1
Record Dates: First submitted 2019-10-30; First posted 2019-11-04 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Adenocarcinoma Metastatic; BRCA1 Mutation; BRCA2 Mutation; Pancreatic Acinar Cell Carcinoma; Pancreatic Ductal Adenocarcinoma; Pancreatic Cancer; Metastatic Pancreatic Cancer; Metastatic Pancreatic Ductal Adenocarcinoma; Breast Cancer Metastatic; Breast Cancer Stage IV; Pancreatic Cancer Stage IV; HER2-negative Breast Cancer; HER2 Negative Breast Carcinoma; Adenocarcinoma of the Breast; PALB2 Gene Mutation; Pancreas Cancer, Metastatic; Pancreas Cancer, Recurrent; Pancreas Cancer; Stage IV Pancreatic Cancer; Stage 4 Pancreatic Cancer
Keywords: pancreatic adenocarcinoma; pancreatic cancer; BRCA; BRCA1; BRCA2; melphalan; BCNU; carmustine; vitamin C; vitamin B12b; autologous stem cell infusion; stage 4 pancreatic cancer; metastatic pancreatic cancer; pancreatic acinar cell carcinoma; pancreatic ductal adenocarcinoma; PDAC; breast cancer; stage 4 breast cancer; stage IV pancreatic cancer; stage IV breast cancer; stem cells; HER2-negative breast cancer; PALB2; metastatic breast cancer; BRCA pancreatic cancer; BRCA breast cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Breast Neoplasms; Neoplasm Metastasis; Recurrence | interventions — Melphalan; Carmustine; Vitamin B 12; Hydroxocobalamin; Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Chemotherapy/stem cell treatment (Experimental)
  Interventions: Drug: Melphalan; Drug: BCNU; Drug: Vitamin B12B; Drug: Vitamin C; Device: Autologous Hematopoietic Stem Cells

INTERVENTIONS:
Drug: Melphalan — Intravenous melphalan (to be given in conjunction with the other listed drugs).
Drug: BCNU — Intravenous BCNU (to be given in conjunction with the other listed drugs).
  Other Names: Carmustine
Drug: Vitamin B12B — Intravenous vitamin B12b (to be given in conjunction with the other listed drugs).
  Other Names: Hydroxocobalamin
Drug: Vitamin C — Intravenous vitamin C (to be given in conjunction with the other listed drugs).
  Other Names: Ascorbic acid, sodium ascorbate
Device: Autologous Hematopoietic Stem Cells — After each cycle of chemotherapy, participants will receive an autologous hematopoietic stem cell infusion.

SUMMARY:
The clinical trial is a phase 1, single-arm trial that will evaluate the safety of the investigational treatment on metastatic pancreatic cancer and metastatic breast cancer. The investigational treatment will involve 2 cycles of a combination of intravenous melphalan, BCNU, vitamin B12b, and vitamin C with autologous hematopoietic stem cell infusion. A dose-escalation schedule is being employed for the vitamin C.

DETAILED DESCRIPTION:
In the current clinical trial, subjects will receive a combination of melphalan, BCNU, vitamin B12b, and vitamin C in conjunction with autologous stem cell infusion. The drug combination is designed to address multiple mechanisms of melphalan resistance.

Investigational Treatment Description:

* Hematopoietic Stem Cell Collection

  1. Granulocyte colony-stimulating factor, and if needed Plerixafor, will be used to mobilize bone marrow stem cells, which will be collected by apheresis.
  2. At least 2 bags of CD34+ cells, each containing at least 2 × 10^6 cells/kg, will be prepared and stored.
  3. Mobilization of hematopoietic stem cells will only occur prior to the first cycle of investigational therapy.
  4. If there is not a sufficient mobilization of stem cells for at least 2 cycles of chemotherapy, then no investigational drugs will be given.
* Investigational Drug Therapy and Stem Cell Infusion

  1. All subjects will receive two cycles of investigational drug therapy with stem cell infusion unless precluded by adverse reactions.
  2. Subjects will receive on day -2:

     1. BCNU
     2. Melphalan
     3. Vitamin B12b
     4. Vitamin C
  3. On day 0, at least 2 × 10^6 CD34+ cells/kg will be infused as per the institution's standard procedures.
  4. Subjects will receive supportive care as per the institution's standard procedures before, during, and after the investigational drug therapy and stem cell infusion.
* Additional Cycles a. Subjects will receive a second cycle of the investigational treatment described immediately above in "Investigational Drug Therapy and Stem Cell Infusion," with an interval of approximately 6 weeks between cycles.

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 18 years.
* Pancreatic or breast cancer, as described below.
* Stage IV (based on AJCC staging guidelines) at the time of enrollment.

  a. Note that potential subjects with stage IV cancer that have had a complete response from prior chemotherapy are still potentially eligible.
* Expected survival time ≥ 6 months, as determined by the investigator.
* Life expectancy not severely limited by diseases other than malignancy, as determined by the investigator.
* Karnofsky score ≥ 60%.
* No chemotherapy within 2 weeks of enrollment.
* Prior surgical resection or ablation of the primary tumor is allowed but not required.
* If post-surgical, the subject must be at least 28 days post-op with the surgical wounds healed and significant complications resolved.
* Potential subjects who have received previous chemotherapy and/or PARP inhibitors may be enrolled.
* Measurable or non-measurable disease by the revised response evaluation criteria in solid tumors (RECIST) v.1.1.
* For potential subjects with a germline BRCA1, BRCA2, or PALB2 mutation:

  a. The mutation must be known to be deleterious or suspected to cause functional impairment as assessed by a CLIA-certified laboratory according to the variant classification criteria described in the study protocol.
* For potential subjects with somatic BRCA1, BRCA2, or PALB2 mutations:

  1. The mutation must be a known or suspected deleterious mutation as assessed by a CLIA-certified laboratory according to the variant classification criteria described in the study protocol.
  2. There must be biallelic loss or inactivation of the mutated BRCA1, BRCA2, or PALB2 gene as assessed by a CLIA-certified laboratory.
  3. The Genetics Review Committee for this trial, which is comprised of a core group of investigators and whose actions are performed in accordance with the committee's charter, must agree that the biallelic mutations are deleterious or suspected deleterious.
* For subjects without a BRCA1, BRCA2, or PALB2 mutation

  1. Subject must have received at least 16 weeks of first-line (platinum-based*) chemotherapy with no evidence of treatment failure, where treatment failure is defined as growing tumors, new lesions, or a steadily rising tumor marker during or within eight weeks of completion of the first line therapy.
  2. * Subjects can also have been treated with FOLFIRINOX but switched to FOLFIRI due to oxaliplatin side effects.
* For potential subjects with pancreatic cancer:

  1. Pancreatic ductal adenocarcinoma or pancreatic acinar cell carcinoma.
  2. If the potential subject has had surgical resection of the primary tumor, then there must be no evidence of disease progression between the time of surgical resection of the primary tumor and screening for enrollment if the patient is seeking enrollment in the immediate post-surgery period.
* For potential subjects with breast cancer:

  1. Adenocarcinoma of the breast.
  2. HER2-negative cancer as per American Society of Clinical Oncology/College of American Pathologists human epidermal growth factor receptor 2 (HER2) testing in breast cancer guidelines.
  3. Male or female sex.
* Histological or cytological confirmation of the primary cancer diagnosis is required.
* Metastatic disease must be histologically or cytologically confirmed unless in the clinical judgment of the investigator a biopsy is not needed for diagnostic purposes.
* Female participants of childbearing potential must agree to do one of the following from the time of signing of the informed consent through 6 months after the last dose of melphalan:

  1. Simultaneously practice two effective barrier methods of contraception. Oral and injectable contraceptives are not allowed. Barrier methods of birth control (e.g., diaphragm and spermicide, or condom and spermicide) are required.
  2. Practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods, and withdrawal) are not acceptable methods of contraception.
* Male participants:

  1. Unless the male is in a monogamous relationship with a female that does not have child-bearing potential, male subjects (even if surgically sterilized) must agree to do one of the following from the time of signing of the informed consent through 6 months after the last dose of melphalan:

     1. Practice effective barrier contraception, plus a second method of effective contraception.
     2. Practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods, and withdrawal) are not acceptable methods of contraception.

Exclusion Criteria

* Rapid disease progression or clinical features concerning for onset of rapid symptomatic deterioration, as determined by the investigator.
* Biliary tract obstruction.
* Current cholangitis. A biliary stent in situ does not otherwise exclude protocol participation.
* A history of only one episode of cholangitis and fewer than 30 days have passed since discontinuation of antibiotic treatment.
* A history of multiple episodes of cholangitis and after discussion between the site study team and sponsor medical monitor and careful evaluation for suitability the patient is deemed to be unsuitable for the trial due to risk of recurring cholangitis.
* Portal hypertension.
* Sinistral portal hypertension.
* Obliteration or significant obstruction of the major veins or arteries (e.g., portal vein, superior mesenteric artery, superior mesenteric vein).
* Clinically significant malignant ascites or malignant pleural effusion, as determined by the investigator.
* Metastatic lesion to the heart or eye.
* Chemotherapy for an indication other than treatment of the current cancer within the past 1 year with a more than 30% risk of recurrence as determined by the investigator.
* Known or suspected metastatic involvement of the central nervous system.
* Left ventricular ejection fraction less than 45% by Multigated Acquisition Scan or echocardiogram (or significantly below the lower limit of normal for the specific test).
* Clinically significant structural heart disease or vascular disease.
* Myocardial infarction within 6 months prior to enrollment; New York Heart Association (NYHA) Class III or IV heart failure; angina; uncontrolled ventricular arrhythmias; or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
* Clinically significant prolongation of QTc (Bazett formula) on EKG, defined as > 0.45 s in males and > 0.47 s in females.
* Severe hypertension, which is defined as the presence of any of the following:

  1. History of hypertensive crisis, hypertensive emergency, or malignant hypertension within the last year.
  2. Sustained or persistent systolic BP > 165 mm Hg or diastolic > 110 mm Hg.
* Other clinically significant cardiovascular disease.
* NOTE:

  1. A past history of severe hypertension that is well-controlled with therapy or that was addressed by removal of the cause (e.g., removal of a medicine that caused the severe hypertension) is not an exclusion criterion.
  2. The presence of a pacemaker is not a contraindication and is not considered an exclusion criterion
* History or evidence of interstitial lung disease (e.g., pneumonitis or pulmonary fibrosis).
* If a smoker, refusal to stop smoking for the duration of the trial.
* FEV1 or DLCO (adjusted for hemoglobin) < 50% of predicted.
* Total bilirubin > 2x upper normal limit, except that potential subjects with Gilbert's Disease are permitted to exceed 2x upper normal limit.
* ALT or AST > 2.5x upper normal limit.
* Alkaline phosphatase > 2.5x upper normal limit, in conjunction with elevated GGT.
* Albumin < 3.0 g/dl.
* Clinical evidence of sinusoidal obstruction syndrome.
* Corrected creatinine clearance consistently < 50 ml/min/1.73 m^2.
* Clinically significant renal disease.
* Hemolytic anemia.
* Family history of catalase deficiency or history or evidence of a severe adverse reaction to hydrogen peroxide consistent with catalase deficiency, unless testing has demonstrated that the patient is not catalase-deficient.
* Evidence of bone marrow insufficiency or failure, in the judgment of the investigator.
* A hemoglobin < 9 g/dL.
* G6PD deficiency as measured by quantitative enzyme levels below the normal reference range in blood.
* Pre-existing bleeding diathesis or coagulopathy.
* Potential subject is pregnant.
* Breast feeding and unwilling to stop.
* Wilson's disease.
* Primary or secondary hemochromatosis.
* Hgb A1c > 9%.
* Hyperuricemia that is not responsive to therapy.
* Plasma oxalate greater than 10 µM, which is not responsive to measures to reduce the level below 10 µM.
* History of clinically significant elevation of plasma oxalic acid or complications related to oxalic acid.
* Prior or current hepatitis B or C.
* HIV infection or seropositivity for HIV.
* Active, clinically significant bacterial, viral, or fungal infection.
* History of colonization with a multidrug-resistant "superbug" that poses a high risk of an untreatable infection in the setting of neutropenia.
* Uncontrolled seizure disorder.
* If a potential subject has received radiation, then any of the following:

  1. A volume ≥ 700 ml of normal liver received a dose ≥ 10 Gy.
  2. The mean dose to normal liver (i.e., liver minus gross tumor volume) was ≥ 10 Gy.
  3. The mean dose to normal lung (i.e., lung minus gross tumor volume) was ≥ 4 Gy.
* History of significant allergy or other contraindication to BCNU, melphalan, vitamin B12b, vitamin C, pegfilgrastim, or Neupogen, or to any excipient in those drugs.
* Use of any of the following cytochrome P450 2b6 (CYP2b6) inducers within 21 days of the planned date of BCNU treatment: phenobarbital, carbamazepam, rifampicin, phenytoin, sulfinpyrazone, or verapamil.
* Disulfiram (Antabuse) use within 30 days of the planned ethanol administration.
* Current chronic use of immunosuppressive agents (e.g., methotrexate, cyclosporine, corticosteroids).
* Prior bone marrow stem cell transplant.
* Except for adjuvant therapy for breast cancer or pancreatic cancer, prior radiation therapy to the brain, kidneys, pelvis, or GI tract or treatment with yttrium-90.
* Prior treatment with bleomycin or BCNU.
* Prior treatment, within 30 days of enrollment, with a drug that has not been FDA-approved for any indication (cancer or otherwise).
* Subject has not fully recovered (i.e., there remain toxicities > Grade 1) from the reversible effects of prior chemotherapy, with the exception of chemotherapy-induced alopecia and grade 2 peripheral neuropathy, unless in the opinion of the principal investigator the effects are not of clinical significance.
* Any concurrent anticancer treatment.
* Serious underlying medical or psychiatric illness or another condition that in the clinical judgment of the principal investigator is likely to interfere with the potential subject completing participation in the trial, based on safety concerns or otherwise.
* Inability or unwillingness to adhere to the study protocol.
* Unwillingness to receive ethanol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-01-13 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Rate of Sinusoidal obstruction syndrome | 30 days after treatment
  Sinusoidal obstruction syndrome diagnosis and grading will use the European Society for Blood and Marrow Transplantation's Revised Diagnosis and Severity Criteria for Sinusoidal Obstruction Syndrome/Veno-Occlusive Disease in Adult Patients as published in 2016. Gradings are from mild to very severe (multi-organ dysfunction/multi-organ failure).
Rate of Idiopathic or Non-Infective Pulmonary Toxicity ≥ Grade 3 | 3 months after the last treatment
  The American Thoracic Society Committee on Idiopathic Pneumonia Syndrome definition will be employed.
Rate of Idiopathic or Non-Infective Pulmonary Toxicity ≥ Grade 3 | 6 months after the last treatment
  The American Thoracic Society Committee on Idiopathic Pneumonia Syndrome definition will be employed.
Rate of Presumptive Oxalate Nephropathy | Within 48 hours of vitamin C treatment
  Oxalate nephropathy will be presumed if there is acute kidney injury or increased creatinine, grade 3 or higher by the criteria of CTCAE Version 5.0 within 48 h of the administration of vitamin C, in the absence of a clear alternative explanation (an example of an alternative explanation is tumor lysis syndrome).
Rate of Cytokine Release Syndrome ≥ Grade 3 | Within 48 hours of each vitamin C treatment
  Cytokine release syndrome will be assessed by the criteria of CTCAE Version 5.0. Elevation of plasma cytokine levels consistent with the diagnosis of cytokine release syndrome must be present.
Rate of Mucositis ≥ Grade 3 | Day 7 after each treatment
  Mucositis will be assessed using the WHO Mucositis Scale. Grading is from 0 (no symptoms) to 4 (no possible alimentation).
Rate of Mucositis ≥ Grade 3 | Day 14 after each treatment
  Mucositis will be assessed using the WHO Mucositis Scale. Grading is from 0 (no symptoms) to 4 (no possible alimentation).
Rate of Mucositis ≥ Grade 3 | Day 21 after each treatment
  Mucositis will be assessed using the WHO Mucositis Scale. Grading is from 0 (no symptoms) to 4 (no possible alimentation).
Rate of Delayed Engraftment of Neutrophils | Day 21 after each treatment
  Neutrophil engraftment is defined as an absolute neutrophil count ≥ 500/microliter for 3 days, with the date of engraftment being the first of those 3 days. Delayed engraftment is engraftment that occurs after 21 days but within 30 days.
Rate of Failed Engraftment of Neutrophils | Day 30 after each treatment
  Neutrophil engraftment is defined as an absolute neutrophil count ≥ 500/microliter for 3 days, with the date of engraftment being the first of those 3 days. Failure to engraft within 30 days will be considered an engraftment failure.
Rate of Delayed Engraftment of Platelets | Day 30 after each treatment
  Platelet engraftment is defined as a platelet count ≥ 20,000/microliter for 3 days, with the date of engraftment being the first of those 3 days. Delayed engraftment is engraftment that occurs after 30 days.
Overall incidence rate of adverse events | Until 12 months after the second stem cell treatment
  Adverse event is defined any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug-related.
Overall incidence rate of serious adverse events | Until 12 months after the second stem cell treatment
  An adverse event is considered serious if, in the view of either the investigator or Sponsor, it results in any of the following outcomes:
  * Death.
  * A life-threatening adverse event.
  * Inpatient hospitalization or prolongation of existing hospitalization.
  * A persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions.
  * A congenital anomaly or birth defect. Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered serious when, based upon appropriate medical judgment, they may jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.
Overall incidence rate of Grade 3-5 adverse events | Until 12 months after the second stem cell treatment
  Grading will be measured using Common Terminology Criteria for Adverse Events version 5.0

SECONDARY OUTCOMES:
Objective response according to RECIST version 1.1 | 1 month after the first stem cell treatment
  Objective response will be evaluated according to RECIST version 1.1 as assessed by the independent core imaging facility. This endpoint will be evaluated with CT scans with contrast of the abdomen, pelvis, and chest and other sites as clinically indicated at each time point.
Objective response according to RECIST version 1.1 | 1 month after the second stem cell treatment
  Objective response will be evaluated according to RECIST version 1.1 as assessed by the independent core imaging facility. This endpoint will be evaluated with CT scans with contrast of the abdomen, pelvis, and chest and other sites as clinically indicated at each time point.
Objective response according to RECIST version 1.1 | 3 months after the second stem cell treatment
  Objective response will be evaluated according to RECIST version 1.1 as assessed by the independent core imaging facility. This endpoint will be evaluated with CT scans with contrast of the abdomen, pelvis, and chest and other sites as clinically indicated at each time point.
Objective response according to RECIST version 1.1 | 6 months after the second stem cell treatment
  Objective response will be evaluated according to RECIST version 1.1 as assessed by the independent core imaging facility. This endpoint will be evaluated with CT scans with contrast of the abdomen, pelvis, and chest and other sites as clinically indicated at each time point.
Objective response according to RECIST version 1.1 | 9 months after the second stem cell treatment
  Objective response will be evaluated according to RECIST version 1.1 as assessed by the independent core imaging facility. This endpoint will be evaluated with CT scans with contrast of the abdomen, pelvis, and chest and other sites as clinically indicated at each time point.
Objective response according to RECIST version 1.1 | 12 months after the second stem cell treatment
  Objective response will be evaluated according to RECIST version 1.1 as assessed by the independent core imaging facility. This endpoint will be evaluated with CT scans with contrast of the abdomen, pelvis, and chest and other sites as clinically indicated at each time point.
Objective response rate in metastatic lesions | 1 month after the first stem cell treatment
  Objective response of metastatic lesions will be evaluated according to RECIST version 1.1 as assessed by the independent core imaging facility, but excluding the primary tumor from the analysis. This endpoint will be evaluated with CT scans with contrast of the abdomen, pelvis, and chest and other sites as clinically indicated at each time point.
Objective response rate in metastatic lesions | 1 month after the second stem cell treatment
  Objective response of metastatic lesions will be evaluated according to RECIST version 1.1 as assessed by the independent core imaging facility, but excluding the primary tumor from the analysis. This endpoint will be evaluated with CT scans with contrast of the abdomen, pelvis, and chest and other sites as clinically indicated at each time point.
Objective response rate in metastatic lesions | 3 months after the second stem cell treatment
  Objective response of metastatic lesions will be evaluated according to RECIST version 1.1 as assessed by the independent core imaging facility, but excluding the primary tumor from the analysis. This endpoint will be evaluated with CT scans with contrast of the abdomen, pelvis, and chest and other sites as clinically indicated at each time point.
Objective response rate in metastatic lesions | 6 months after the second stem cell treatment
  Objective response of metastatic lesions will be evaluated according to RECIST version 1.1 as assessed by the independent core imaging facility, but excluding the primary tumor from the analysis. This endpoint will be evaluated with CT scans with contrast of the abdomen, pelvis, and chest and other sites as clinically indicated at each time point.
Objective response rate in metastatic lesions | 9 months after the second stem cell treatment
  Objective response of metastatic lesions will be evaluated according to RECIST version 1.1 as assessed by the independent core imaging facility, but excluding the primary tumor from the analysis. This endpoint will be evaluated with CT scans with contrast of the abdomen, pelvis, and chest and other sites as clinically indicated at each time point.
Objective response rate in metastatic lesions | 12 months after the second stem cell treatment
  Objective response of metastatic lesions will be evaluated according to RECIST version 1.1 as assessed by the independent core imaging facility, but excluding the primary tumor from the analysis. This endpoint will be evaluated with CT scans with contrast of the abdomen, pelvis, and chest and other sites as clinically indicated at each time point.
Overall Survival | Until 12 months after the second stem cell treatment
  Overall survival will be measured from the time of enrollment until death from any cause and will be measured in the intent-to-treat population. Subjects without a known date of death will be censored on the date the subject was last known to be alive.
Progression-Free Survival | Until 12 months after the second stem cell treatment
  Progression-free survival will be measured as time-to-progression with the starting time being the time of enrollment.
  A subject is also considered to have progressed if one of the following occurs:
  * Progression as determined by a RECIST evaluation.
  * Unequivocal evidence of clinical progression.
  * Marked escalation in cancer-related pain that is assessed by the principal investigator to indicate the need for other systemic chemotherapy.
  * Immediate need for initiation of new anticancer treatment or surgical or radiological intervention for complications due to tumor progression even in the absence of radiological progression.
  * Marked deterioration in Karnofsky score felt by the investigator to indicate clinical progression.
  * A determination that it is in the best interest of the subject to come off the study due to clinical progression.
  * Death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Arnold Glazier, M.D., Study Director — General Oncology, Inc.
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York